CLINICAL TRIAL: NCT07261111
Title: Effect of Subtle Energy Transmission and Tao Calligraphy Mindfulness Practice on Mitochondrial DNA (mtDNA) in Peripheral Blood Leukocytes
Brief Title: Effect of Subtle Energy Transmission and Tao Calligraphy Mindfulness Practice on Mitochondrial DNA in Peripheral Blood Leukocytes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sha Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00090526
Record Dates: First submitted 2025-11-21; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Mitochondrial DNA; Quality of Life
Keywords: Mitochondrial-to-nuclear genome ratio; Tao Calligraphy; Mindfulness Practice; Healing Art; Healing Song; Meditation; SF-36 Questionnaire; Mitochondrial DNA; Mitochondrial DNA content; Quality of life

STUDY DESIGN:
Intervention Model Description: We plan subjects may enter the study as a group and will have all measurements (blood sample for Mitochondrial DNA analysis and Rand SF 36 Questionnaire) done upon entry into the study - at the baseline 0-time point; at the 3-months time point, at the 6-months time point and at the 12-months time point.
  Participants will start practices at baseline time point and will stop practices at 12-months time-point.
  The study will evaluate the effects of mindfulness practice using:
  * The standardized Quality of Life SF-36 Questionnaire.
  * Mitochondrial DNA content in peripheral blood Leukocytes. All participants will have blood drawn and complete the questionnaire upon entry into the study - Baseline time point; at 3-months time point, at six-months time point and at twelve-months time point.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The Practice Group (Experimental): The Practice group will start practices at baseline time-point and will stop practices after 12 months at 12-months time-point. The participants in Practice group will practice Mindfulness practice with Calligraphy at least 30 minutes daily for 12 months. All participants in Practice group will have the blood drawn for Mitochondrial DNA content analysis and complete the SF-36 questionnaire upon entry into the study - Baseline time-point; at 3-months time-point, at six-months time point and at twelve-months time point.
  Interventions: Other: Mindfulness practice with Tao Art (Calligraphy and Song Greatest Love)

INTERVENTIONS:
Other: Mindfulness practice with Tao Art (Calligraphy and Song Greatest Love) — During mindfulness practice with Tao Art (Calligraphy and Greatest Love Song), participants will repeatedly trace the lines of calligraphy with fingers while listening to, singing, or chanting with Tao Song. This enables them to achieve deep concentration, while maintaining fully alert state. The practice can be done in sitting or standing, depending on the health status and age and will last 30 minutes and is done daily for 12 months.

SUMMARY:
The goal of this pilot clinical trial is to learn if a subtle energy transmission and Tao Calligraphy Mindfulness Practice works to improve mitochondrial DNA. The main questions it aims to answer are:

* Does Tao Calligraphy Mindfulness practice improve mitochondrial DNA content in peripheral blood leucocytes in adults?
* Will this improvement of mitochondrial DNA content in peripheral blood leucocytes be statistically significant? Researchers will compare the values of mitochondrial DNA content in peripheral blood leucocytes at beginning of the mindfulness practices to the values at 3 months, 6 months and 12 months of practice group.

Participants will:

* have blood samples will drawn at accredited institutions and analyzed for Mitochondrial DNA content in Leucocytes upon entry into the study - Baseline time point; at 3-months time point, at six-months time point and at twelve-months time point.
* All participants will complete the set of 3 questionnaires upon entry into the study - Baseline time point; at 3-months time point, at six-months time point and at twelve-months time point.
* Practice the Mindfulness with Tao Calligraphy minimum 30 minutes daily.

DETAILED DESCRIPTION:
Objective

The goal of this study is to measure the effects of a unique form of Tao Calligraphy mindfulness practice that involves engaging with Tao art (tracing the Tao Calligraphy "Greatest Love" while listening to or singing the Tao Music or Tao Song "Greatest Love") together with subtle energy transmission on Mitochondrial DNA in peripheral blood leucocytes.

In our previous study, the participants who regularly practiced, shown an increase of the length in telomeres in peripheral blood granulocytes. In our other studies, participants reported a decrease in symptoms of their illness as perceived subjectively, improved signs reported by treating clinicians and an improvement of well-being as measured by standardized scientific questionnaires.

Hypotheses

The research null hypothesis is that individuals who receive subtle energy transmission for mitochondrial DNA in hemato-lymphoid tissue, and who will engage in daily Tao Calligraphy mindfulness practice for 12 months, will have no significant change in Mitochondrial DNA content in peripheral blood leucocytes in follow-up analyses and will show no improvement of well-being as measured by standardized scientific questionnaire Rand SF-36 at 3, 6 and 12 months.

For statistical analysis of the data from laboratory assessment and scores obtained from questionnaires, the Anova, T-Test and regression analysis will be used to evaluate the null hypothesis. The p value will represent how unlikely the observed data would be if the null hypothesis were actually true and investigators will use them to reach conclusions. The confidence level is set at 95% and if we receive p < 0.05, then H0 is rejected. The correlation coefficient will be used to determine any correlation between various factors (e.g. effects of age, sex, length, and frequency of mindfulness practices and other) on outcome and regression analysis will be used to determine the relation of independent and dependent variables.

Tools such as the Minitabs version 14 and or Statistical Package for the Social Sciences (SPSS) or Free version of Statistical Package for the Social Sciences (PSPP) will be used.

Background and Theoretical Framework

Mitochondria are membrane bound, self-replicating organelles present in almost all eukaryotic cells. Mitochondrial energy production is essential for all cellular processes. In general, each human cell contains several hundred to 1,000 mitochondria, each with 2-10 copies of Mitochondrial DNA encoding 13 proteins essential for respiratory chain function. Thought to have originated from symbiotic ancestors, mitochondria contribute to many processes central to cellular function and dysfunction including calcium signalling, cell growth and differentiation, cell cycle control and cell death. Mitochondrial shape and positioning in cells is tightly regulated by processes of fission and fusion, biogenesis and autophagy, ensuring a relatively constant mitochondrial population. Mitochondrial inheritance is generally accepted to be maternal although small amounts of paternally transmitted mitochondria have been discovered on rare occasions.

Mitochondrial dysfunction is considered one of the hallmarks of aging and age-associated diseases. The mitochondrial genome is more vulnerable to oxidative damage and undergoes a higher rate of mutation compared with nuclear DNA. Additional underlying causes of mitochondrial dysfunction include inadequate mitochondrial quantity, exposure to environmental toxins, reduction in mitochondrial membrane permeability, impaired transport of essential metabolites, and malfunctioning of the electron transport chain and Adenosine triphosphate (ATP) synthesis.

Unfortunately, no measure is currently available that globally assesses the ability of mitochondria to perform normal biological functions. Mitochondrial functions include but are not limited to oxidative phosphorylation and energy production in the form of Adenosine triphosphate (ATP) , reactive oxygen species (ROS) production, cell death signalling, as well as steroid hormone synthesis, and systemic signalling.

It has been proposed that the number of Mitochondrial DNA copies per cell (Mitochondrial DNA copy number) reflects mitochondrial health. A major driver of the popularity of Mitochondrial DNA copy number as a potential marker of mitochondrial health lies in its ease of measure from stored DNA, or indirectly from genotyping/sequencing data. Compared to direct assays of mitochondrial function, which require fresh tissue, the scalability of Mitochondrial DNA copy number assessments is appealing for biomarker studies.

However, Mitochondrial DNA copy number does not directly reflect respiratory chain (RC) function or energy production capacity. According to the theory of "biochemical threshold", only when Mitochondrial DNA copy number decreases by 60 to 80% of normal levels does RC function and energy production capacity decrease. This means that in many cases 20-40% of the baseline Mitochondrial DNA copy number is sufficient to produce the 13 proteins necessary to sustain respiratory capacity. But this level of Mitochondrial DNA depletion seems to occur only in rare mitochondrial diseases or in isolated single cells in diseased organs. The uncoupling of Mitochondrial DNA copy number and respiratory capacity may be accounted for by the fact that up-regulation of transcription and translation from pre-existing Mitochondrial DNA copies can increase the levels of messenger ribonucleic acid (mRNA), protein subunits, RC function, and energy production capacity, without a change in Mitochondrial DNA copy number. This notably occurs in response to exercise, where mitochondrial content and RC activity in human muscle increases within days to weeks without a change in Mitochondrial DNA copy number. Thus, in human tissues, Mitochondrial DNA copy number is not directly coupled to, and does not directly reflect mitochondrial bioenergetics.

Furthermore, the picture is somewhat complicated in that while low blood Mitochondrial DNA copy number has been associated with neurodegenerative disease, cardiovascular disease, and both cognitive and physical performance in aging; other conditions such as diabetes, major depression, some cancers, and mitochondrial disorders are associated with elevated Mitochondrial DNA copy number. Regarding exposure to environmental toxicants, Mitochondrial DNA copy number has been associated with either higher or lower Mitochondrial DNA copy number.

Nevertheless, the value and specificity of blood Mitochondrial DNA copy number can be increased in several ways as summarized below:

1. Use data from complete blood counts with differential, enhanced using flow cytometry methods that quantify immunologically-defined cell subpopulations, then analyses with multivariate models (i.e., deconvolution method) to understand the proportion of variance in Mitochondrial DNA copy number attributable not just to general immune cell categories (e.g., granulocytes and lymphocytes) but to specific cell subtypes (naive and memory cluster of differentiation 4 (CD4) and cluster of differentiation 8 (CD8) T cells, B cells, subtypes of monocytes, etc).
2. Further enhance the sensitivity and interpretability of Mitochondrial DNA copy number in relation to health related phenotypes by quantifying Mitochondrial DNA copy number directly in molecularly-defined subtypes of immune cells. For example, CD4+ Naive T cells, monocytes, or other specific immune subtype exist in sufficient abundance in circulation to be isolated by either flow cytometric cell sorting (also known as fluorescence-activated cell sorting, FACS) or by negative/positive selection by magnetic activated cell sorting. Compared to cell mixtures, cell-specific Mitochondrial DNA copy number quantification add biological specificity to detect meaningful mitochondrial associations related to exposures, other biomarkers, and possibly age and sex-related differences.
3. Measure other markers of mitochondrial content and/or function in parallel with Mitochondrial DNA copy number, e.g. live assays of mitochondrial function. Some examples include i) citrate synthase (CS) activity, cardiolipin, or mitochondrial protein abundance to estimate mitochondrial content; ii) Mitochondrial DNA integrity, such as DNA damage, point mutations, or deletions; or iii) mitochondrial respiratory capacity, such as oxygen consumption by respirometry, which can and should be performed in specific cell types, as well as respiratory chain enzymatic activities that reflect energy production capacity on either a per-cell or per-mitochondrion basis. In the context of direct measurements of respiratory chain function, Mitochondrial DNA copy number becomes a more biologically interpretable feature of mitochondrial health.
4. Measure circulating markers of mitochondrial stress accessible in plasma or other bio fluids, including Growth Differentiation Factor 15 (GDF15), cf Mitochondrial DNA or other emerging mitochondrial kinesis. However, these may lack specificity. E.g. GDF15, cf Mitochondrial DNA, and other circulating markers can be induced by a number of stressors not necessarily reflecting mitochondrial RC capacity or stress.
5. There is a negative correlation between the copy number of Mitochondrial DNA, number of mutations in mitochondrial deoxyribonucleic acid (Mitochondrial DNA) and longevity. Higher rates of somatic Mitochondrial DNA mutations are consistently associated with aging phenotypes, increased risk of age-related diseases, and reduced lifespan in both animal models and human populations.
6. Whole Mitochondrial DNA sequencing (via next-generation sequencing or Sanger sequencing) can identify single nucleotide polymorphisms (SNPs), haplogroups, and mutational burden associated with longevity. This approach enables detection of specific SNPs and haplogroups that have been associated with increased lifespan.
7. The mitochondrial-to-nuclear genome ratio (Mitochondrial DNA content) in tissues and body fluids correlates with the size and number of mitochondria. Polymerase Chain Reaction (PCR) based molecular test to determine mitochondrial-to-nuclear genome ratio in peripheral blood leukocytes.

It has been concluded that although the biological interpretation of differences in Mitochondrial DNA copy number is tenuous, in combination with relevant markers assessed in homogenous or well-defined cell populations, continuing to add Mitochondrial DNA copy number to existing studies with rich sets of outcomes is likely to contribute valuable insights into the role of mitochondria in human health, aging, and resilience.

Mindfulness Practices and Mitochondria

Psychologically, mindfulness reduces cognitive and emotional reactivity, rumination, and worry, while increasing self-awareness and acceptance, which mediate improvements in mental health and facilitate healthier behaviours. These psychological changes are tightly linked to the observed biological effects.

The biological mechanisms by which mindfulness practices improve health involve down-regulation of stress and inflammatory pathways, enhancement of immune function, and neoplastic changes supporting self-regulation and adaptive coping.

Mindfulness practices may contribute to prolonging human life by improving mitochondrial function, reducing cellular stress, and promoting adaptive stress responses that enhance cellular maintenance and resilience. Chronic psychological stress accelerates mitochondrial dysfunction, increases oxidative damage, and impairs cellular repair mechanisms, all of which are associated with aging and reduced lifespan. Mindfulness-based interventions have been shown to mitigate these effects by reducing stress-induced inflammation and oxidative stress, thereby supporting mitochondrial health.

Mitochondria regulate key longevity pathways through energy production, redox signalling, and mitochondrial-nuclear communication. Mindfulness practices can activate beneficial mitochondrial stress responses, such as mitochondrial hormesis, which involves mild mitochondrial stress that triggers adaptive cellular repair and maintenance mechanisms, ultimately promoting longevity in animal models and potentially in humans. These responses include enhanced osteoporosis, increased expression of overprotective factors, and improved metabolic efficiency.

Chinese calligraphy

Chinese calligraphy handwriting is a dynamic process of integrating visual spatial awareness, cognitive planning and motor skills that is maneuvered with a brush to follow defined configurations of characters. There have been growing empirical studies of Chinese calligraphic handwriting that resulted in improvements in visual attention and span, increased mental concentration, confirming it as an effective treatment for psychosomatic conditions and post-traumatic hyper-arousal symptoms and exhibited significant effects on hypertension and type 2 diabetes. Leisure activities occurring later in life that includes calligraphy may inhibit cognitive decline.

Tao Calligraphy is a unique branch of Chinese calligraphy (Yi Bi Zi) in that it is characterized by one-stroke writing. Every character is written with one continuous stroke with the brush always in contact with the paper. Results from studies confirmed efficacy in tracing in post-acute rehabilitation setting in that patients reported less incontinence, shortened duration of hospital stay, and an increase in overall well-being. Retrospective analysis of data exhibited improvement in general wellbeing, an increase in optimism and energy level, as well as improvement of their symptoms. According to a study measuring the effects of calligraphy tracing meditation with mantra chanting (repeated sound or word to aid with concentration spoken out loud or silently) of spiritual practitioners, the results exhibited statistically positive improvement in Physical Functioning, Role Limitations due to physical health problems; Role Limitations due to Personal or Emotional Problems; Energy / Fatigue; Emotional Well-being; Social Functioning; Bodily Pain; General Health. In the prospective follow up study of these subjects, following 6 months they continued to improve in functioning in the above-mentioned areas. The authors concluded that tracing calligraphy and mantra chanting was simple to follow, well tolerated, and no complications arose during the study.

The investigators have already discussed the value of Tao art mindfulness meditations for improving depression, anxiety, pain, cancer and health, length of Telomeres in Leucocytes and how this appears to contribute to beneficial outcomes related to well-being (Quality of Life score SF-36).

ELIGIBILITY:
Inclusion Criteria:

* Age 19 and over
* Willingness and ability to comply with data collection requirements
* Submission of required documentation before entering the study, including informed consent and consent to release of information
* Healthy or Ill, with the exception of genetic illnesses and cancer (for which treatments could negatively impact measurement) and serious mental disorders (e.g. bipolar disorder, schizophrenia, psychosis),
* Willingness to allow their data to be used for research purposes and published as deemed fit (while conforming to all applicable privacy laws) by Sha Research Foundation.
* Willingness to practice the daily calligraphy meditations and follow the protocol.

Exclusion Criteria:

* Not meeting any of the inclusion criteria
* Bipolar disorders, other serious mental disorders (e.g. schizophrenia, psychosis), genetic illnesses (primarily affected chromosomes), and cancer (treatment could negatively impact telomere during research period)
* inability to sign consent and follow instructions
* Unwillingness to participate in data gathering
* Unable to follow the practice regimen, including the daily calligraphy meditations
* Pregnant or nursing. Participants who become pregnant during the study will be required to end their participation. (to avoid any, at current time unknown, potential negative effect of the study on the fetus).
* There are no exclusion criteria placed upon potential subjects related to national origin, culture, ethnicity, race, sex, physical disability, sexual orientation, religion, or spiritual practices.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-02 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean Change from Baseline in Mitochondrial-to-nuclear genome ratio (Mitochondrial DNA content) in peripheral blood Leukocytes at 3 months, 6 months and 12 months | From start of Mindfulness practices with Tao Art (Calligraphy and Song Greatest Love) to end of practices at 12 months
  Genomic DNA is extracted from peripheral blood and DNA concentration and purity are assessed by spectrophotometer. Mitochondrial DNA content in leukocytes is quantified by real-time quantitative PCR. Calculating Mitochondrial DNA content is done as follows: Ct values for Mitochondrial DNA targets are normalized to the nuclear gene Ct using the delta-delta cycle threshold method, using equation: Mitochondrial DNA content = relative Mitochondrial DNA abundance / nuclear DNA abundance. This ratio reflects the relative number of mitochondrial genomes per nuclear genome in leukocytes.
  The normal range for the mitochondrial-to-nuclear genome ratio (Mitochondrial DNA/ Nuclear DNA) in human blood leukocytes is approximately 1.2 to 1.8.

SECONDARY OUTCOMES:
Mean Change from Baseline in Quality of Life Scores on 36-item short-form Quality of Life Questionnaire (SF-36) at 3 months, 6 months and 12 months | From start of Mindfulness practices with Tao Art (Calligraphy and Song Greatest Love) to end of practices at 12 months.
  A 36-item short-form Quality of Life Questionnaire (SF-36) was constructed to survey health status. The investigators chose the longer 36-item version to assess the impact of the Tao art mindfulness practice and drinking energized water on Quality of Life of participants with unipolar depression.
  The SF-36 includes one multi-item scale for eight health concepts:
  1. limitations in physical activities;
  2. limitations in social activities;
  3. limitations in usual role activities;
  4. bodily pain;
  5. general mental health (psychological distress and well-being);
  6. limitations in usual role activities because of emotional problems;
  7. vitality (energy and fatigue);
  8. general health perceptions. Through a complex calculation, eight scores are derived from answers to 36 questions of SF-36. Finally, these eight scores are linearly transformed to a 0-to-100 scale, with 100 being the best possible outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hudoba De Badyn, MD, FRCS, Principal Investigator — Sha Research Foundation; Cynthia Hamilton, PhD, Principal Investigator — Sha Research Foundation
Locations (1):
- Sha Research Foundation (BC Branch), North Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
Investigators will share the change in the mean of the mitochondrial-to-nuclear genome ratio (Mitochondrial DNA content) in peripheral blood leucocytes in follow-up analyses and the change in the mean score of SF-36 questionnaire after 12 months of Mindfulness Practices with Tao Art. These will be posted to Clinical trials website at completion of study December 31 2031 and will be available until December 31 2032.
Supporting Information: Study Protocol, SAP
Time Frame: Investigators will share the protocol of the study upon acceptance to Clinical trials website by December 31 2025. It will be available until end of the study December 31 2031.
Access Criteria: Anyone with active account with Clinical trials website will be able to access the Individual Participant Data (IPD) and supporting information. They will be able to access Protocol, statistical plan and mean score of all 3 questionnaires. They will be able to access it through Clinical trials website platform.

REFERENCES:
- [Background] Patin E, Hasan M, Bergstedt J, Rouilly V, Libri V, Urrutia A, Alanio C, Scepanovic P, Hammer C, Jonsson F, Beitz B, Quach H, Lim YW, Hunkapiller J, Zepeda M, Green C, Piasecka B, Leloup C, Rogge L, Huetz F, Peguillet I, Lantz O, Fontes M, Di Santo JP, Thomas S, Fellay J, Duffy D, Quintana-Murci L, Albert ML; Milieu Interieur Consortium. Natural variation in the parameters of innate immune cells is preferentially driven by genetic factors. Nat Immunol. 2018 Mar;19(3):302-314. doi: 10.1038/s41590-018-0049-7. Epub 2018 Feb 23. PMID 29476184
- [Result] Osellame LD, Blacker TS, Duchen MR. Cellular and molecular mechanisms of mitochondrial function. Best Pract Res Clin Endocrinol Metab. 2012 Dec;26(6):711-23. doi: 10.1016/j.beem.2012.05.003. Epub 2012 Jun 23. PMID 23168274
- [Result] Knez J, Winckelmans E, Plusquin M, Thijs L, Cauwenberghs N, Gu Y, Staessen JA, Nawrot TS, Kuznetsova T. Correlates of Peripheral Blood Mitochondrial DNA Content in a General Population. Am J Epidemiol. 2016 Jan 15;183(2):138-46. doi: 10.1093/aje/kwv175. Epub 2015 Dec 24. PMID 26702630
- [Result] Trumpff C, Michelson J, Lagranha CJ, Taleon V, Karan KR, Sturm G, Lindqvist D, Fernstrom J, Moser D, Kaufman BA, Picard M. Stress and circulating cell-free mitochondrial DNA: A systematic review of human studies, physiological considerations, and technical recommendations. Mitochondrion. 2021 Jul;59:225-245. doi: 10.1016/j.mito.2021.04.002. Epub 2021 Apr 9. PMID 33839318
- [Result] de Witte M, Orkibi H, Zarate R, Karkou V, Sajnani N, Malhotra B, Ho RTH, Kaimal G, Baker FA, Koch SC. From Therapeutic Factors to Mechanisms of Change in the Creative Arts Therapies: A Scoping Review. Front Psychol. 2021 Jul 15;12:678397. doi: 10.3389/fpsyg.2021.678397. eCollection 2021. PMID 34366998
- [Result] Marikar Bawa FL, Mercer SW, Sutton JW, Bond CM. Mindfulness for people with chronic pain: Factors affecting engagement and suggestions for programme optimisation. Health Expect. 2023 Jun;26(3):1287-1307. doi: 10.1111/hex.13745. Epub 2023 Mar 12. PMID 36908018
- [Result] Wallace DC. The epigenome and the mitochondrion: bioenergetics and the environment [corrected]. Genes Dev. 2010 Aug 1;24(15):1571-3. doi: 10.1101/gad.1960210. PMID 20679390
- [Result] O'Hara R, Tedone E, Ludlow A, Huang E, Arosio B, Mari D, Shay JW. Quantitative mitochondrial DNA copy number determination using droplet digital PCR with single-cell resolution. Genome Res. 2019 Nov;29(11):1878-1888. doi: 10.1101/gr.250480.119. Epub 2019 Sep 23. PMID 31548359
- [Result] Picard M, Wallace DC, Burelle Y. The rise of mitochondria in medicine. Mitochondrion. 2016 Sep;30:105-16. doi: 10.1016/j.mito.2016.07.003. Epub 2016 Jul 14. PMID 27423788
- [Result] Picard M. Blood mitochondrial DNA copy number: What are we counting? Mitochondrion. 2021 Sep;60:1-11. doi: 10.1016/j.mito.2021.06.010. Epub 2021 Jun 19. PMID 34157430
- [Result] White JD. National Cancer Institute's support of research to further integrative oncology practice. J Natl Cancer Inst Monogr. 2014 Nov;2014(50):286-7. doi: 10.1093/jncimonographs/lgu036. No abstract available. PMID 25749590
- [Result] Jamil A, Gutlapalli SD, Ali M, Oble MJP, Sonia SN, George S, Shahi SR, Ali Z, Abaza A, Mohammed L. Meditation and Its Mental and Physical Health Benefits in 2023. Cureus. 2023 Jun 19;15(6):e40650. doi: 10.7759/cureus.40650. eCollection 2023 Jun. PMID 37476142
- [Result] Lan Q, Lim U, Liu CS, Weinstein SJ, Chanock S, Bonner MR, Virtamo J, Albanes D, Rothman N. A prospective study of mitochondrial DNA copy number and risk of non-Hodgkin lymphoma. Blood. 2008 Nov 15;112(10):4247-9. doi: 10.1182/blood-2008-05-157974. Epub 2008 Aug 18. PMID 18711000
- [Result] Gardi C, Fazia T, Stringa B, Giommi F. A short Mindfulness retreat can improve biological markers of stress and inflammation. Psychoneuroendocrinology. 2022 Jan;135:105579. doi: 10.1016/j.psyneuen.2021.105579. Epub 2021 Nov 6. PMID 34775250
- [Result] Roubicek DA, Souza-Pinto NC. Mitochondria and mitochondrial DNA as relevant targets for environmental contaminants. Toxicology. 2017 Nov 1;391:100-108. doi: 10.1016/j.tox.2017.06.012. Epub 2017 Jun 26. PMID 28655544
- [Result] Rossignol R, Faustin B, Rocher C, Malgat M, Mazat JP, Letellier T. Mitochondrial threshold effects. Biochem J. 2003 Mar 15;370(Pt 3):751-62. doi: 10.1042/BJ20021594. PMID 12467494
- [Result] Puente-Maestu L, Lazaro A, Tejedor A, Camano S, Fuentes M, Cuervo M, Navarro BO, Agusti A. Effects of exercise on mitochondrial DNA content in skeletal muscle of patients with COPD. Thorax. 2011 Feb;66(2):121-7. doi: 10.1136/thx.2010.153031. Epub 2010 Nov 20. PMID 21097816
- [Result] Pahal S, Mainali N, Balasubramaniam M, Shmookler Reis RJ, Ayyadevara S. Mitochondria in aging and age-associated diseases. Mitochondrion. 2025 May;82:102022. doi: 10.1016/j.mito.2025.102022. Epub 2025 Feb 27. PMID 40023438
- [Result] Osto C, Benador IY, Ngo J, Liesa M, Stiles L, Acin-Perez R, Shirihai OS. Measuring Mitochondrial Respiration in Previously Frozen Biological Samples. Curr Protoc Cell Biol. 2020 Dec;89(1):e116. doi: 10.1002/cpcb.116. PMID 33320426
- [Result] Meyer JN, Hartman JH, Mello DF. Mitochondrial Toxicity. Toxicol Sci. 2018 Mar 1;162(1):15-23. doi: 10.1093/toxsci/kfy008. PMID 29340618
- [Result] Lopez-Otin C, Blasco MA, Partridge L, Serrano M, Kroemer G. Hallmarks of aging: An expanding universe. Cell. 2023 Jan 19;186(2):243-278. doi: 10.1016/j.cell.2022.11.001. Epub 2023 Jan 3. PMID 36599349
- [Result] De Valois RL. Contribution of different lateral geniculate cell types to visual behavior. Vision Res. 1971;Suppl 3:383-96. doi: 10.1016/0042-6989(71)90052-6. No abstract available. PMID 5293880
- [Result] Kim C, Bassig BA, Seow WJ, Hu W, Purdue MP, Huang WY, Liu CS, Cheng WL, Mannisto S, Vermeulen R, Weinstein SJ, Lim U, Hosgood HD, Bonner MR, Caporaso NE, Albanes D, Lan Q, Rothman N. Mitochondrial DNA copy number and chronic lymphocytic leukemia/small lymphocytic lymphoma risk in two prospective studies. Cancer Epidemiol Biomarkers Prev. 2015 Jan;24(1):148-53. doi: 10.1158/1055-9965.EPI-14-0753. Epub 2014 Oct 7. PMID 25293880
- [Result] Hu W, Zhang J, Wu Z, Wu Y, Hu Y, Hu X, Cao J. Research progress on paternal mitochondrial inheritance: An overview. Mitochondrion. 2025 May;82:102019. doi: 10.1016/j.mito.2025.102019. Epub 2025 Feb 28. PMID 40024491
- [Result] Grunewald A, Rygiel KA, Hepplewhite PD, Morris CM, Picard M, Turnbull DM. Mitochondrial DNA Depletion in Respiratory Chain-Deficient Parkinson Disease Neurons. Ann Neurol. 2016 Mar;79(3):366-78. doi: 10.1002/ana.24571. Epub 2016 Jan 28. PMID 26605748
- [Result] Forsstrom S, Jackson CB, Carroll CJ, Kuronen M, Pirinen E, Pradhan S, Marmyleva A, Auranen M, Kleine IM, Khan NA, Roivainen A, Marjamaki P, Liljenback H, Wang L, Battersby BJ, Richter U, Velagapudi V, Nikkanen J, Euro L, Suomalainen A. Fibroblast Growth Factor 21 Drives Dynamics of Local and Systemic Stress Responses in Mitochondrial Myopathy with mtDNA Deletions. Cell Metab. 2019 Dec 3;30(6):1040-1054.e7. doi: 10.1016/j.cmet.2019.08.019. Epub 2019 Sep 12. PMID 31523008
- [Result] Egan B, O'Connor PL, Zierath JR, O'Gorman DJ. Time course analysis reveals gene-specific transcript and protein kinetics of adaptation to short-term aerobic exercise training in human skeletal muscle. PLoS One. 2013 Sep 12;8(9):e74098. doi: 10.1371/journal.pone.0074098. eCollection 2013. PMID 24069271
- [Result] Copeland WC, Wachsman JT, Johnson FM, Penta JS. Mitochondrial DNA alterations in cancer. Cancer Invest. 2002;20(4):557-69. doi: 10.1081/cnv-120002155. PMID 12094550
- [Result] Cai N, Chang S, Li Y, Li Q, Hu J, Liang J, Song L, Kretzschmar W, Gan X, Nicod J, Rivera M, Deng H, Du B, Li K, Sang W, Gao J, Gao S, Ha B, Ho HY, Hu C, Hu J, Hu Z, Huang G, Jiang G, Jiang T, Jin W, Li G, Li K, Li Y, Li Y, Li Y, Lin YT, Liu L, Liu T, Liu Y, Liu Y, Lu Y, Lv L, Meng H, Qian P, Sang H, Shen J, Shi J, Sun J, Tao M, Wang G, Wang G, Wang J, Wang L, Wang X, Wang X, Yang H, Yang L, Yin Y, Zhang J, Zhang K, Sun N, Zhang W, Zhang X, Zhang Z, Zhong H, Breen G, Wang J, Marchini J, Chen Y, Xu Q, Xu X, Mott R, Huang GJ, Kendler K, Flint J. Molecular signatures of major depression. Curr Biol. 2015 May 4;25(9):1146-56. doi: 10.1016/j.cub.2015.03.008. Epub 2015 Apr 23. PMID 25913401
- [Result] Boulet L, Karpati G, Shoubridge EA. Distribution and threshold expression of the tRNA(Lys) mutation in skeletal muscle of patients with myoclonic epilepsy and ragged-red fibers (MERRF). Am J Hum Genet. 1992 Dec;51(6):1187-200. PMID 1334369
- [Result] Ashar FN, Zhang Y, Longchamps RJ, Lane J, Moes A, Grove ML, Mychaleckyj JC, Taylor KD, Coresh J, Rotter JI, Boerwinkle E, Pankratz N, Guallar E, Arking DE. Association of Mitochondrial DNA Copy Number With Cardiovascular Disease. JAMA Cardiol. 2017 Nov 1;2(11):1247-1255. doi: 10.1001/jamacardio.2017.3683. PMID 29049454
- [Result] Zhang D, Lee EKP, Mak ECW, Ho CY, Wong SYS. Mindfulness-based interventions: an overall review. Br Med Bull. 2021 Jun 10;138(1):41-57. doi: 10.1093/bmb/ldab005. PMID 33884400
- [Result] Kao H Sr, Zhu L, Chao AA, Chen HY, Liu IC, Zhang M. Calligraphy and meditation for stress reduction: an experimental comparison. Psychol Res Behav Manag. 2014 Feb 13;7:47-52. doi: 10.2147/PRBM.S55743. eCollection 2014. PMID 24611024
- [Result] Bugugnani MJ, Leroy G, Richard L, Haiat R. [Lipid evaluation can be performed within the 1st 24 hours after myocardial infarction]. Presse Med. 1986 Jun 28;15(26):1217-8. No abstract available. French. PMID 2944090

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-09-30): https://cdn.clinicaltrials.gov/large-docs/11/NCT07261111/Prot_SAP_000.pdf